CLINICAL TRIAL: NCT05824767
Title: DPP3, Angiotensin II, and Renin Kinetics in Sepsis (DARK-Sepsis) Pilot: Serum Biomarkers to Predict Response to Angiotensin II vs. Standard-of-care Vasopressor Therapy in the Treatment of Septic Shock, a Randomized Controlled Pilot Trial
Brief Title: Serum Biomarkers to Predict Response to Angiotensin II in Septic Shock
Acronym: DARK-Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Principal Investigator, Joao P. Teixeira, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-111
Record Dates: First submitted 2023-03-05; First posted 2023-04-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Septic Shock; Vasodilatory Shock
Keywords: septic shock; vasopressor; angiotensin II; renin; dipeptidyl peptidase 3 (DPP3); randomized controlled trial
MeSH Terms: conditions — Shock, Septic | interventions — Angiotensin II; Giapreza

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Angiotensin II (Experimental): For patients randomized to the intervention group, once the dose of background norepinephrine reaches ≥0.10 mcg/kg/min for ≥30 minutes, angiotensin II will be started at a dose of 20 ng/kg/min (recommended starting dose in package insert).Thereafter, angiotensin II and norepinephrine will both be titrated to mean arterial pressure (MAP) goal of >/= 65 mmHg according to the protocol titration scheme and in accordance with the University of New Mexico Hospital (UNMH) Nursing Department Titration Guideline. Angiotensin II treatment will be capped at 72 hours, at which point (if a second vasopressor is still needed) the patient will be started on an alternative agent.
  Interventions: Drug: Angiotensin II
- Standard of Care (SOC) (No Intervention): Vasopressor therapy be titrated by the clinical team per usual SOC and UNMH Nursing Department Titration Guideline. using other available vasopressor agents (e.g., higher-dose norepinephrine, vasopressin, epinephrine, phenylephrine, and/or dopamine). To provide a comparator arm, patients in the SOC will have renin and DPP3 levels obtained at equivalent timepoints.

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II (Giapreza) is a pharmacologic version of a naturally occurring peptide hormone of the same name which is a component of the renin-angiotensin-aldosterone system (RAAS). Angiotensin II (Giapreza) was FDA-approved in 2017 as a vasoconstrictive agent in the treatment of vasodilatory shock.
  Other Names: Giapreza
  Arms: Angiotensin II

SUMMARY:
This trial will be a randomized controlled single-center pilot trial comparing the use of angiotensin II versus standard-of-care (SOC) vasopressor therapy in adult patients with persistent vasodilatory shock despite moderate-dose norepinephrine, with a primary outcome of the ability of novel biomarkers (renin and DPP3) to predict blood pressure response to angiotensin II. Given our angiotensin II will be compared to SOC, this will be an unblinded study.

DETAILED DESCRIPTION:
Sepsis affects >1 million Americans yearly and, when septic shock ensues, it is associated with high morbidity and mortality. Though first-line norepinephrine is standard of care, there are limited prospective data to guide the choice of additional vasopressors in septic shock. While more studies are needed, preliminary data suggest that the vasopressor angiotensin II (AngII) may improve outcomes in septic shock, especially in certain subsets of patients, such as those with acute kidney injury (AKI) requiring renal replacement therapy (RRT), acute respiratory distress syndrome (ARDS), or high severity of illness.

Furthermore, there are no validated biomarkers currently available to guide the choice of vasopressor therapy in septic shock. In this study the investigators will evaluate two potential biomarkers, renin and dipeptidyl peptidase 3 (DPP3). Renin has been shown in preliminary studies to accurately predict mortality in septic shock, outperforming lactate, and to predict beneficial response to AngII. A less well-known candidate biomarker is DPP3, which is an aminopeptidase that cleaves a variety of biologically active oligopeptides including angiotensin II. Similar to renin, preliminary observational data show that elevated DPP3 levels in patients with sepsis are associated with organ dysfunction and short-term mortality, outperforming lactate as a predictor of death.

This study is an unblinded pilot randomized controlled trial (RCT) comparing AngII (intervention) to standard-of-care (SOC) vasopressor therapy in adult patients with persistent vasodilatory shock requiring moderate dose norepinephrine. The primary outcome will be the ability of renin and DPP3 to predict blood pressure (BP) response to AngII. As both renin and DPP3 are associated with overall short-term prognosis in sepsis, the SOC arm will allow us to determine if the predictive value of renin and DPP3 is specific to AngII therapy. A variety of secondary clinical outcomes will also be tracked, but the primary purpose of this pilot study is to inform the future design of a large multicenter RCT evaluating the biomarker-guided use of angiotensin II as a second-line vasopressor in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years-old with persistent vasodilatory shock despite moderate-dose norepinephrine monotherapy, defined as those who require ≥0.1 mcg/kg/min for at least 30 minutes to maintain a MAP between 65-70 mmHg.
* Patients are required to have central venous and arterial catheters present, and they are expected to remain in place for at least the initial 72 hours of study.
* Patients are required to have an indwelling urinary catheter present, and it is expected to remain in place for at least the 72 hours of study.
* Patients must have received 20-30 mL/kg of crystalloid over the previous 24-hour period, as clinically appropriate, and no longer be fluid responsive as per UNMH protocol. By UNMH protocol, lack of fluid responsiveness is considered a failure to increase stroke volume, stroke volume index, cardiac output, or cardiac index (typically measured by non-calibrated pulse contour analysis using a FloTrac device) by at least 10% after a 500-mL crystalloid bolus or a passive leg raise. Patients for whom the treating physicians feel that 20 mL/kg of crystalloid may be clinically inappropriate can qualify for the study if the reason for withholding further IV fluids is documented.
* Patient or (in patients unable to consent) legal authorized representative (LAR) is willing and able to provide written informed consent and comply with all protocol requirements.
* Approval from the attending physician and clinical pharmacist conducting the study.

Exclusion Criteria:

* Patients who are < 18 years of age.
* Patients diagnosed with acute occlusive coronary syndrome requiring intervention and/or cardiogenic shock.
* Patients with or suspected to have abdominal aortic aneurysm or aortic dissection.
* Acute stroke.
* Patients with acute mesenteric ischemia or those with a history of mesenteric ischemia.
* Patients with known Raynaud's phenomenon, systemic sclerosis, or vasospastic disease.
* Patients on venoarterial extracorporeal membrane oxygenation (VA-ECMO).
* Patients with liver failure with a Model for End-Stage Liver Disease (MELD) score of =/>30.
* Patients with burns covering >20% of total body surface area.
* Patients with a history of asthma or chronic obstructive pulmonary disease (COPD) with active acute bronchospasm or (if not mechanically ventilated) with an acute exacerbation of their asthma/COPD requiring the use of inhaled bronchodilators.
* Patients requiring more than 500 mg daily of hydrocortisone or equivalent glucocorticoid medication as a standing dose.
* Patients with an absolute neutrophil count (ANC) of < 1,000/mm3
* Patients with hemorrhagic shock OR active bleeding AND an anticipated need (within 48 hours of initiation of the study) for transfusion of >4 units of packed red blood cells.
* Patients with active bleeding AND hemoglobin < 7g/dL or any other condition that would contraindicate serial blood sampling.
* Untreated venous thromboembolism (VTE) or inability to tolerate pharmacologic VTE prophylaxis.
* Patients with a known allergy to mannitol.
* Patients with an expected survival of <24 hours, SOFA score ≥ 16, or death deemed to be imminent or inevitable during the admission.
* Either the attending physician or patient and/or substitute decisionmaker are not committed to all active treatment, e.g., do-not-resuscitate (DNR) status.
* Patients who are known to be pregnant at the time of screening. All women ≤50 years-old will need a negative serum pregnancy test (serum quantitative beta-hCG) to enroll.
* Prisoner status
* Patients who are currently participating in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Ability of baseline renin to predict norepinephrine equivalent dose (NED) at 3 hours | 3 hours post drug initiation or SOC equivalent
  BP response will be assessed at 3 hours in both groups and measured using NED. The primary outcome will be ability of baseline renin (obtained at drug initiation or equivalent SOC timepoint) to predict total NED at 3 hours, using treatment arm (AngII vs. SOC) and baseline Sequential Organ Failure Assessment (SOFA) scores as covariables.
Ability of baseline DPP3 to predict NED at 3 hours | 3 hours post drug initiation or SOC equivalent
  BP response will be assessed at 3 hours in both groups and measured using NED. The primary outcome will be ability of baseline DPP3 to predict total NED at 3 hours, using treatment arm (AngII vs. SOC) and baseline SOFA scores as covariables.

SECONDARY OUTCOMES:
Ability of pre-baseline renin to predict NED at 3 hours | 3 hours post drug initiation or SOC equivalent
  The primary outcome analysis will be repeated, but instead using the ability of pre-baseline renin levels (obtained at randomization, approximately 2 hours before drug initiation or equivalent SOC timepoint) to predict total NED at 3 hours, using treatment arm (AngII vs. SOC) and baseline SOFA scores as covariables.
Ability of pre-baseline DPP3 to predict NED at 3 hours | 3 hours post drug initiation or SOC equivalent
  The primary outcome analysis will be repeated, but instead using the ability of pre-baseline DPP3 levels (obtained at randomization, approximately 2 hours before drug initiation or equivalent SOC timepoint) to predict total NED at 3 hours, using treatment arm (AngII vs. SOC) and baseline SOFA scores as covariables.
Ability of changes in renin level to predict NED at 3 hours | 3 hours post drug initiation or SOC equivalent
  The primary outcome analysis will be repeated, but instead evaluating the ability of changes in renin level (from pre-baseline to baseline) to predict total NED at 3 hours, using treatment arm (AngII vs. SOC) and baseline SOFA scores as covariables.
Ability of changes in DPP3 level to predict NED at 3 hours | 3 hours post drug initiation or SOC equivalent
  The primary outcome analysis will be repeated, but instead evaluating the ability of changes in DPP3 level (from pre-baseline to baseline) to predict total NED at 3 hours, using treatment arm (AngII vs. SOC) and baseline SOFA scores as covariables.
Background NED at 1 hour | 1 hour post drug initiation or SOC equivalent
  Comparison of background NED in AngII arm and SOC arm will be compared at multiple timepoints.
Background NED at 6 hours | 6 hours post drug initiation or SOC equivalent
  Comparison of background NED in AngII arm and SOC arm will be compared at multiple timepoints.
Background NED at 12 hours | 12 hours post drug initiation or SOC equivalent
  Comparison of background NED in AngII arm and SOC arm will be compared at multiple timepoints.
Background NED at 24 hours | 24 hours post drug initiation or SOC equivalent
  Comparison of background NED in AngII arm and SOC arm will be compared at multiple timepoints.
Background NED at 48 hours | 48 hours post drug initiation or SOC equivalent
  Comparison of background NED in AngII arm and SOC arm will be compared at multiple timepoints.
Background NED at 72 hours | 72 hours post drug initiation or SOC equivalent
  Comparison of background NED in AngII arm and SOC arm will be compared at multiple timepoints.
Time to shock reversal | 72 hours post drug initiation or SOC equivalent
  Time (in hours) to sustained vasopressor independence will be compared in two arms.
Change in Sequential Organ Failure Assessment (SOFA) score at 24 hours | 24 hours post drug initiation or SOC equivalent
  Change in SOFA score from baseline to 24 hours. (SOFA score ranges from 0 to 24, with higher score indicating worse organ function.)
Change in Sequential Organ Failure Assessment (SOFA) score at 48 hours | 48 hours post drug initiation or SOC equivalent
  Change in SOFA score from baseline to 24 hours. (SOFA score ranges from 0 to 24, with higher score indicating worse organ function.)
Change in Sequential Organ Failure Assessment (SOFA) score at 72 hours | 72 hours post drug initiation or SOC equivalent
  Change in SOFA score from baseline to 24 hours. (SOFA score ranges from 0 to 24, with higher score indicating worse organ function.)
Acute Kidney Injury (AKI) | 28 days post randomization
  Rate of AKI during first 28 days as defined by KDIGO (Kidney Disease: Improving Global Outcomes) criteria
Days free from renal replacement therapy (RRT) | 28 days post randomization
  Days alive and free from RRT. Freedom from RRT is considered a period without RRT of at least 72 hours. Specified as a key secondary outcome.
Days free from invasive mechanical ventilation (IMV) | 28 days post randomization
  Days alive and free from IMV. Specified as a key secondary outcome.
Intensive care unit (ICU) length of stay | Until ICU discharge or study termination, up to 26 weeks.
  Length of stay (in days)
Hospital length of stay | Until hospital discharge or study termination, up to 26 weeks.
  Length of stay (in days)
ICU mortality | Until ICU discharge or 28 days post-randomization.
  Death before ICU discharge. Specified as a key secondary outcome.
Hospital mortality | Until hospital discharge or 28 days post-randomization.
  Death before hospital discharge. Specified as a key secondary outcome.

OTHER OUTCOMES:
serum renin level at 1 hour | 1 hour post-drug initiation and SOC equivalent
  To generate a deeper understanding of renin kinetics, renin levels will be obtained at multiple equivalent timepoints in both arms, with approximately 2 hours between randomization and AngII initiation in the AngII arm.
serum DPP3 level at 1 hour | 1 hour post-drug initiation and SOC equivalent
  To generate a deeper understanding of DPP3 kinetics, DPP3 levels will be obtained at multiple equivalent timepoints in both arms, with approximately 2 hours between randomization and AngII initiation in the AngII arm.
serum renin level at 3 hours | 3 hours post-drug initiation and SOC equivalent
  To generate a deeper understanding of renin kinetics, renin levels will be obtained at multiple equivalent timepoints in both arms, with approximately 2 hours between randomization and AngII initiation in the AngII arm.
serum DPP3 level at 3 hours | 3 hours post-drug initiation and SOC equivalent
  To generate a deeper understanding of DPP3 kinetics, DPP3 levels will be obtained at multiple equivalent timepoints in both arms, with approximately 2 hours between randomization and AngII initiation in the AngII arm.
serum renin level at 24 hours | 24 hours post-drug initiation and SOC equivalent
  To generate a deeper understanding of renin kinetics, renin levels will be obtained at multiple equivalent timepoints in both arms, with approximately 2 hours between randomization and AngII initiation in the AngII arm.
serum DPP3 level at 24 hours | 24 hours post-drug initiation and SOC equivalent
  To generate a deeper understanding of DPP3 kinetics, DPP3 levels will be obtained at multiple equivalent timepoints in both arms, with approximately 2 hours between randomization and AngII initiation in the AngII arm.
serum renin level 24 hours post drug discontinuation | 24 hours post-drug discontinuation (AngII arm only)
  To evaluate for a rebound effect, final biomarker levels will be obtained in the AngII arm at approximately 24 hours after drug discontinuation.
serum DPP3 level 24 hours post drug discontinuation | 24 hours post-drug discontinuation (AngII arm only)
  To evaluate for a rebound effect, final biomarker levels will be obtained in the AngII arm at approximately 24 hours after drug discontinuation.
Prespecified Adverse Events: new venous thromboembolism (VTE) or arterial thrombosis | Up to 28 days
  Requires radiographic documentation. For events to be considered adverse events (AEs) they must be new hospital-acquired events which developed after randomization.
Prespecified Adverse Events: atrial fibrillation | Up to 28 days
  For events to be considered adverse events (AEs) they must be new hospital-acquired events which developed after randomization.
Prespecified Adverse Events: tachycardia | Up to 28 days
  Tachycardia is defined as new rise in heart rate to >100/min sustained for at least 1 hour.
  For events to be considered adverse events (AEs) they must be new hospital-acquired events which developed after randomization.
Prespecified Adverse Events: lactic acidosis | Up to 28 days
  Defined as rise in serum lactate level to above the upper limit of normal. For lactic acidosis to be considered an adverse event, lactate level must be higher than pre-randomization level.
Prespecified Adverse Events: hyperglycemia | Up to 28 days
  Defined as rise in blood glucose level to above the upper limit of normal. For hyperglycemia to be considered an adverse event, glucose level must be higher than pre-randomization level.
Prespecified Adverse Events: thrombocytopenia | Up to 28 days
  Defined as drop in platelet count to below the lower limit of normal. For thrombocytopenia to be considered an adverse event, the platelet level must be lower than pre-randomization level.
Prespecified Adverse Events: peripheral limb/digit ischemia | Up to 28 days
  As diagnosed by clinical team. For events to be considered adverse events (AEs) they must be new hospital-acquired events which developed after randomization.
Prespecified Adverse Events: intestinal ischemia | Up to 28 days
  As diagnosed by clinical team. For events to be considered adverse events (AEs) they must be new hospital-acquired events which developed after randomization.
Prespecified Adverse Events: confirmed infection | Up to 28 days
  Requires the infecting organism to be confirmed by culture or other identification method; administration of appropriate antimicrobial therapy (if available); and clinical documentation of infection. For events to be considered adverse events (AEs) they must be new hospital-acquired events which developed after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Joao P Teixeira, MD, Principal Investigator — University of New Mexico; Nathan D Nielsen, MD MSc, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
Reasonable requests for data will be considered on a case-by-case basis and will require regulatory approval by both University of New Mexico and the study sponsor (La Jolla Pharmaceutical).

REFERENCES:
- [Background] Teixeira JP, Perez Ingles D, Barton JB, Dean JT, Garcia P, Kunkel SJ, Sarangarm P, Weiss NK, Schaich CL, Busse LW, Nielsen ND. The scientific rationale and study protocol for the DPP3, Angiotensin II, and Renin Kinetics in Sepsis (DARK-Sepsis) randomized controlled trial: serum biomarkers to predict response to angiotensin II versus standard-of-care vasopressor therapy in the treatment of septic shock. Trials. 2024 Mar 12;25(1):182. doi: 10.1186/s13063-024-07995-0. PMID 38475822
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Background] Tumlin JA, Murugan R, Deane AM, Ostermann M, Busse LW, Ham KR, Kashani K, Szerlip HM, Prowle JR, Bihorac A, Finkel KW, Zarbock A, Forni LG, Lynch SJ, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Bellomo R; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Outcomes in Patients with Vasodilatory Shock and Renal Replacement Therapy Treated with Intravenous Angiotensin II. Crit Care Med. 2018 Jun;46(6):949-957. doi: 10.1097/CCM.0000000000003092. PMID 29509568
- [Background] Gordon AC, Mason AJ, Thirunavukkarasu N, Perkins GD, Cecconi M, Cepkova M, Pogson DG, Aya HD, Anjum A, Frazier GJ, Santhakumaran S, Ashby D, Brett SJ; VANISH Investigators. Effect of Early Vasopressin vs Norepinephrine on Kidney Failure in Patients With Septic Shock: The VANISH Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):509-18. doi: 10.1001/jama.2016.10485. PMID 27483065
- [Background] Gleeson PJ, Crippa IA, Mongkolpun W, Cavicchi FZ, Van Meerhaeghe T, Brimioulle S, Taccone FS, Vincent JL, Creteur J. Renin as a Marker of Tissue-Perfusion and Prognosis in Critically Ill Patients. Crit Care Med. 2019 Feb;47(2):152-158. doi: 10.1097/CCM.0000000000003544. PMID 30653055
- [Background] Bellomo R, Forni LG, Busse LW, McCurdy MT, Ham KR, Boldt DW, Hastbacka J, Khanna AK, Albertson TE, Tumlin J, Storey K, Handisides D, Tidmarsh GF, Chawla LS, Ostermann M. Renin and Survival in Patients Given Angiotensin II for Catecholamine-Resistant Vasodilatory Shock. A Clinical Trial. Am J Respir Crit Care Med. 2020 Nov 1;202(9):1253-1261. doi: 10.1164/rccm.201911-2172OC. PMID 32609011
- [Background] Busse L, Albertson T, Gong M. Outcomes in patients with acute respiratory distress syndrome receiving angiotensin II for vasodilatory shock [Abstract P125]. Crit Care.2018;22(Suppl 1):82 (50).
- [Background] Nguyen M, Denimal D, Dargent A, Guinot PG, Duvillard L, Quenot JP, Bouhemad B. Plasma Renin Concentration is Associated With Hemodynamic Deficiency and Adverse Renal Outcome in Septic Shock. Shock. 2019 Oct;52(4):e22-e30. doi: 10.1097/SHK.0000000000001285. PMID 30407370
- [Background] Kullmar M, Saadat-Gilani K, Weiss R, Massoth C, Lagan A, Cortes MN, Gerss J, Chawla LS, Fliser D, Meersch M, Zarbock A. Kinetic Changes of Plasma Renin Concentrations Predict Acute Kidney Injury in Cardiac Surgery Patients. Am J Respir Crit Care Med. 2021 May 1;203(9):1119-1126. doi: 10.1164/rccm.202005-2050OC. PMID 33320784
- [Background] Flannery AH, Ortiz-Soriano V, Li X, Gianella FG, Toto RD, Moe OW, Devarajan P, Goldstein SL, Neyra JA. Serum renin and major adverse kidney events in critically ill patients: a multicenter prospective study. Crit Care. 2021 Aug 14;25(1):294. doi: 10.1186/s13054-021-03725-z. PMID 34391450
- [Background] Jeyaraju M, McCurdy MT, Levine AR, Devarajan P, Mazzeffi MA, Mullins KE, Reif M, Yim DN, Parrino C, Lankford AS, Chow JH. Renin Kinetics Are Superior to Lactate Kinetics for Predicting In-Hospital Mortality in Hypotensive Critically Ill Patients. Crit Care Med. 2022 Jan 1;50(1):50-60. doi: 10.1097/CCM.0000000000005143. PMID 34166293
- [Background] Meersch M, Weiss R, Massoth C, Kullmar M, Saadat-Gilani K, Busen M, Chawla L, Landoni G, Bellomo R, Gerss J, Zarbock A. The Association Between Angiotensin II and Renin Kinetics in Patients After Cardiac Surgery. Anesth Analg. 2022 May 1;134(5):1002-1009. doi: 10.1213/ANE.0000000000005953. PMID 35171852
- [Background] Deniau B, Blet A, Santos K, Vaittinada Ayar P, Genest M, Kastorf M, Sadoune M, de Sousa Jorge A, Samuel JL, Vodovar N, Bergmann A, Mebazaa A, Azibani F. Inhibition of circulating dipeptidyl-peptidase 3 restores cardiac function in a sepsis-induced model in rats: A proof of concept study. PLoS One. 2020 Aug 27;15(8):e0238039. doi: 10.1371/journal.pone.0238039. eCollection 2020. PMID 32853284
- [Background] Rehfeld L, Funk E, Jha S, Macheroux P, Melander O, Bergmann A. Novel Methods for the Quantification of Dipeptidyl Peptidase 3 (DPP3) Concentration and Activity in Human Blood Samples. J Appl Lab Med. 2019 May;3(6):943-953. doi: 10.1373/jalm.2018.027995. Epub 2018 Nov 30. PMID 31639686
- [Background] Blet A, Deniau B, Santos K, van Lier DPT, Azibani F, Wittebole X, Chousterman BG, Gayat E, Hartmann O, Struck J, Bergmann A, Antonelli M, Beishuizen A, Constantin JM, Damoisel C, Deye N, Di Somma S, Dugernier T, Francois B, Gaudry S, Huberlant V, Lascarrou JB, Marx G, Mercier E, Oueslati H, Pickkers P, Sonneville R, Legrand M, Laterre PF, Mebazaa A; AdrenOSS-1 Study Investigators. Monitoring circulating dipeptidyl peptidase 3 (DPP3) predicts improvement of organ failure and survival in sepsis: a prospective observational multinational study. Crit Care. 2021 Feb 15;25(1):61. doi: 10.1186/s13054-021-03471-2. PMID 33588925
- [Background] Picod A, Deniau B, Vaittinada Ayar P, Genest M, Julian N, Azibani F, Mebazaa A. Alteration of the Renin-Angiotensin-Aldosterone System in Shock: Role of the Dipeptidyl Peptidase 3. Am J Respir Crit Care Med. 2021 Feb 15;203(4):526-527. doi: 10.1164/rccm.202010-3873LE. No abstract available. PMID 33152252
- [Background] Jentzer JC, Vallabhajosyula S, Khanna AK, Chawla LS, Busse LW, Kashani KB. Management of Refractory Vasodilatory Shock. Chest. 2018 Aug;154(2):416-426. doi: 10.1016/j.chest.2017.12.021. Epub 2018 Jan 9. PMID 29329694
- [Background] Goradia S, Sardaneh AA, Narayan SW, Penm J, Patanwala AE. Vasopressor dose equivalence: A scoping review and suggested formula. J Crit Care. 2021 Feb;61:233-240. doi: 10.1016/j.jcrc.2020.11.002. Epub 2020 Nov 14. PMID 33220576